CLINICAL TRIAL: NCT01300416
Title: Open, Multi-centre, Non-interventional, Observational Study to Characterize the Impact That GI Complaints Have on Patient-reported Outcomes in Patients Who Have Had a Renal Transplant. Patients Will be Evaluated at Visit 1 and Then Again After 4 (+2) Weeks (Visit 2)
Brief Title: Measurement of Patient Reported Outcomes in Renal Transplant Patients With And Without Gastrointestinal (GI) Symptoms
Acronym: PROGIS
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CERL080AMY02
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Kidney Transplantation; GI Symptoms Severity
Keywords: Kidney transplantation; mycophenolate sodium; EC-MPS; Health Related Quality of Life; GI symptoms; Immunosuppressants; HRQL; PGWB; GIQLI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With Gastro-Intestinal (GI) symptoms
- Without GI symptoms

SUMMARY:
This study will access the GI complaints on patients reported outcomes and to determine the improvement in quality of life in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient received kidney transplant at least 1 month prior to study with MMF as a part of the treatment for at least 2 weeks.
* Eligible to convert to myfortic because of GI complaints or not currently experiencing GI complaints and stable on current immunosuppressive regimen.
* At least 18 years of age;
* Willing to provide written informed consent; and
* Able to meet all study requirements including completing paper questionnaires and completing two study visits.

Exclusion Criteria:

* GI symptoms assumed or known not be caused by MPA therapy and have recent acute rejection at least 1 week prior to the study.
* Breast-feeding or pregnant woman.
* Patients with psychiatric illness.
* Underlying acute medical intervention or hospitalization
* Receiving investigational drug within 30days prior to study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplanted Patients currently on MMF who have GI symptoms and will be converted to EC-MPS treatment and patients currently on MMF without GI symptoms who will continue with MMF therapy.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To determine if GI symptoms severity and health related quality of life of patients has improved after being converted from MMF to EC-MPS due to GI complaints. | 4-6 weeks

SECONDARY OUTCOMES:
To identify and evaluate quality of life and impact on symptom severity based on patients perception. | 4-6 weeks

CONTACTS AND LOCATIONS:
Locations (9):
- Malaysia (9):
  - Hospital Universiti Kebangsaan Malaysia, Cheras
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - Hospital Queen Elizabeth, Kota Kinabalu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Umum Sarawak, Kuching
  - Hospital Pulau Pinang, Pulau Pinang
  - Hospital Selayang, Selayang Baru Utara
  - Hospital Serdang, Serdang